CLINICAL TRIAL: NCT05958524
Title: Analysis of Factors Influencing the Efficacy of Levamlodipine Benzoate and Its Population Pharmacodynamic Modeling
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-49
Record Dates: First submitted 2023-06-02; First posted 2023-07-24 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-08

CONDITIONS: Hypertensive Patients; Monotherapy
Keywords: levamlodipine besylate；monotherapy；; Population pharmacodynamics

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. Preliminarily explore the correlation factors of differences in the efficacy of levamlodipine besylate in the treatment of hypertension.
2. Quantitatively analyze the influence of covariates such as patient demographic factors, personal history, combined medications, and biochemical indicators on the efficacy of levamlodipine besylate, and establish a population pharmacokinetic model of levamlodipine besylate, to achieve clinical Individualized treatment and rational drug use.

DETAILED DESCRIPTION:
This study is a retrospective study, which intends to collect and extract relevant information from outpatient medical records from the information center of our hospital, and evaluate the difference in the efficacy of antihypertensive treatment with levamlodipine besylate in newly diagnosed hypertensive patients in our hospital; After antihypertensive treatment with levamlodipine besylate, the correlation analysis was carried out on the influencing factors of blood pressure control in the follow-up, and the covariates such as demographic factors, personal history, combined medications, and biochemical indicators were initially explored. The curative effect of dipine.

Through the population pharmacokinetic modeling method of quantitative pharmacology, the influence of covariates such as demographic factors, personal history, combined medication, and biochemical indicators on the curative effect of levamlodipine besylate was quantitatively explored. The population pharmacokinetic model of levamlodipine besylate was established in order to provide reference for clinical individualized treatment and rational drug use.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed patients with hypertension in our hospital (sex, age is not limited).
2. Patients whose initial treatment is levamlodipine besylate.

Exclusion Criteria:

1. Patients who cannot be followed up regularly or are lost to follow-up after initial diagnosis and treatment.
2. Patients who were initially treated with other antihypertensive drugs.
3. Blood pressure was not measured when the patient came to the hospital for follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed hypertension who were treated with levamlodipine besylate tablets.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
The systolic blood pressure | Patient's follow-up after initial treatment was 1 month
  The systolic blood pressure was measured at rest
The diastolic blood pressure | Patient's follow-up after initial treatment was 1 month
  The diastolic blood pressure was measured at rest

CONTACTS AND LOCATIONS:
Overall Officials: Xian Yu, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- Yu Xian, Chongqing, China

IPD SHARING:
Plan to Share IPD: No